CLINICAL TRIAL: NCT03263039
Title: Biomarker Discovery Study to Identify Patients With Advanced Urothelial Cancer Benefitting From Pembrolizumab Treatment
Brief Title: Biomarkers in Urothelial Cancer Patients Treated With Pembrolizumab
Acronym: RESPONDER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, M.P.J.K. Lolkema, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL61719.056.17
Record Dates: First submitted 2017-08-18; First posted 2017-08-28 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Transitional Cell Carcinoma of the Bladder; Biomarkers
Keywords: Programmed Cell Death 1 Receptor; Pembrolizumab; Keytruda; MK-3475; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with pembrolizumab (Other): Pembrolizumab will be administered at a flat dose of 200 mg as a 30 minute (-5 min/+10 min) IV infusion every 3 weeks (Q3W)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg Q3W
  Other Names: MK-3475; Keytruda

SUMMARY:
In the RESPONDER study, the role of the immune evasive mechanisms combined with genomic characterization will be explored in urothelial cancer patients treated with second-line treatment with pembrolizumab.

Combined profiling of immune and molecular status is novel and may contribute to improved patient stratification and provide rationale for future treatment strategies containing pembrolizumab.

DETAILED DESCRIPTION:
Antibodies that target the crosstalk between immune and cancer cells by inhibiting programmed death 1 (PD-1, Pembrolizumab and Durvalumab) or programmed death-ligand 1 (PD-L1, Atezolizumab) have shown promising results as second-line treatments in phase II studies with response rates of about 30%.

Although urothelial cancer is prone to immune checkpoint blockade, better understanding of the underlying mechanisms is necessary to improve patient selection. The efficacy of immune checkpoint inhibitors in urothelial cancer may be affected by both tumor specific and environmental factors. In order to improve the efficacy of immunotherapy in urothelial cancer, drivers of local immune suppression need to be identified.

In this prospective translational multicenter study, clinical data, peripheral blood and sequential tumor biopsies are collected from urothelial cancer patients treated with second-line treatment with pembrolizumab to identify the role of immune evasive mechanisms combined with genomic characterization. A pre-treatment tumor biopsy and blood sample will be obtained and subsequently whole genome sequencing and whole genome RNA sequencing is performed. Both tumor tissue as well as peripheral blood will be investigated for immune and molecular profiling. A biopsy will also be taken after start of treatment (at 6 weeks) and at progression (optional)

For future research projects, longitudinal blood samples will be collected for isolation of immune cells, cytokine/chemo-attractants and circulating tumor DNA (ctDNA).

ELIGIBILITY:
Inclusion Criteria:

1. Should have signed informed consent for CPCT-02 (this is another clinical trial, NCT01855477)
2. Be willing and able to provide written informed consent for the trial.
3. Be >= 18 years of age on day of signing informed consent.
4. Have histologically or cytologically-confirmed urothelial cancer that is not amenable to curative treatment with local and/or systemic therapies.
5. Have progressive disease after platinum containing chemotherapy as defined by:

   1. Disease progression after treatment with a platinum-containing regimen for recurrent (disease not amenable to curative treatment)/metastatic disease
   2. Recurrence/progression within 12 months of prior therapy containing platinum
6. Have measurable disease based on RECIST 1.1. Tumor lesions located in a previously irradiated area are considered measurable if progression has been demonstrated in these lesions.
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
8. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
9. Demonstrate adequate organ function according to screening labs, which should be performed within 10 days of treatment initiation.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. lf the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in protocol - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in protocol- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Treatment with an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving high dose systemic steroid therapy (defined as >=; 20 mg prednisone or equivalent per day) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Tuberculosis Bacillus).
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., :S Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., :S Grade 1 or at baseline) from adverse events due to a previously administered agent

   * Note: Subjects with Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using high dose steroids (defined as >=; 20 mg prednisone or equivalent per day) for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subjects participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the prescreening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L 1, or anti- PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has a known history ofor is positive for hepatitis B (hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (hepatitis C virus [HCV] RNA [qualitative] is detected). Note: Without known history, testing needs to be performed to determine eligibility.

    Hepatitis C antibody (Ab) testing is allowed for screening purposes in countries where HCV RNA is not part of standard of care.
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2022-08-19 (Estimated); Study Completion 2023-08-19 (Estimated)

PRIMARY OUTCOMES:
Biomarkers in patients with clinical benefit | End of study (pembrolizumab will be given for a maximum of 24 months), which is within 3 years after start of inclusion
  Peripheral blood and sequential tumor biopsies are collected before start of treatment, during treatment, and (optionally) at progression.
  Immune profiling using in situ multiplex immunofluorescence will be performed to identify tumor epithelial and stromal cells, effector immune cells, T cell co-inhibition, T cell recruitment and immune-suppressive cells. Furthermore, serum samples will be assessed for levels of cytokines/chemoattractants. Finally, longitudinal blood samples will be collected for isolation of immune cells, cytokine/chemo-attractants and ctDNA.
  A qualified pathologist will determine tumor cell percentage in the obtained biopsies. DNA will be obtained from both cancer cells (biopsy tissue) and normal white blood cells (peripheral blood) and will be submitted for whole genome sequencing.
  The obtained data will contribute to identifying potential biomarkers in patients with clinical benefit.

SECONDARY OUTCOMES:
Mechanisms of primary and acquired resistance to pembrolizumab | End of study (pembrolizumab will be given for a maximum of 24 months), which is anticipated to be within 3 years after start inclusion.
  Combined profiling of immune and molecular status (as described in outcome 1) during treatment and at disease progression will reveal different mechanisms by which urothelial cancer evades pembrolizumab.
  Additional bio-informatic analyses will be done to detect the somatic structural variants and copy number changes. The genome data will be used to explore potential correlations between specific pathway aberrations, total number of somatic variants and pattern of mutational load characteristic of the DNA mutational agent and clinical outcome. Moreover, we will perform whole genome RNA sequencing, an essential part of the genomic analysis to identify tumor specific neo-antigens.
  The obtained data will contribute to identifying mechanisms of primary and acquired resistance to pembrolizumab.
Correlations between biomarkers and clinical activity | End of study (pembrolizumab will be given for a maximum of 24 months), which is anticipated to be within 3 years after start inclusion.
  The following definitions and response evaluation criteria will be used to assess potential correlation: immune related response criteria (irRC), duration of response according to RECIST and irRC, duration of clinical benefit (CR-complete response/PR-partial response/SD-stable disease) according to RECIST and irRC, progression-free survival, and overall survival.
  By combining the data from the profiling of immune and molecular status (as described in outcome 1) with the additional data from bio-informatic analyses (as described in outcome 2) and the clinical activity (as described above), correlations between biomarkers and clinical activity can be identified.

OTHER OUTCOMES:
Translation experiments | Collection of samples will be until end of study (pembrolizumab will be given for a maximum of 24 months), which is anticipated to be within 3 years after start inclusion.
  To collect tissue, blood and urine samples for future translational experiments

CONTACTS AND LOCATIONS:
Overall Officials: M.P.J.K. Lolkema, Principal Investigator — Erasmus Medical Center; A.A.M. van der Veldt, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Information can be shared by importing it into another databases

REFERENCES:
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306